CLINICAL TRIAL: NCT01981395
Title: A Double Blind, Randomized, Placebo Controlled, Crossover Study to Investigate the Anti-hyperalgesic Efficacy of a Single Dose of Fenobam on Heat/Capsaicin Induced Cutaneous Hyperalgesia in Adult Healthy Volunteers.
Brief Title: Fenobam on Heat/Capsaicin Induced Hyperalgesia in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laura Cavallone (Other)
Responsible Party: Sponsor-Investigator, Laura Cavallone, Assistant Professor of Anesthesiology, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 201311094
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Hyperalgesia; Allodynia
Keywords: fenobam; heat; capsaicin; hyperalgesia; allodynia; mood; cognitive function
MeSH Terms: conditions — Hyperalgesia | interventions — fenobam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment regimn 1 (Experimental): 150 mg Fenobam Orally - once
  Interventions: Drug: Fenobam
- Treatment Regimen 2 (Placebo Comparator): Placebo orally - once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenobam — Fenobam 150 mg will be administered and subjects will be monitored for up to 8 hours. During the study day questionnaires will be administered, blood will be drawn a testing site will be marked and pain testing and heat/capsaicin sensitization will be measured.
  Other Names: [1-(3-chlorophenyl)-3-(1-methyl-4-oxo-2-imidazolidinylidine) urea hydrate]
  Arms: Treatment regimn 1
Drug: Placebo — A placebo will be administered and subjects will be monitored for up to 8 hours. During the study day questionnaires will be administered, blood will be drawn a testing site will be marked and pain testing and heat/capsaicin sensitization will be measured.
  Other Names: Lactose monohydrate
  Arms: Treatment Regimen 2

SUMMARY:
Our goal is to demonstrate that healthy volunteers treated with fenobam will develop a significantly reduced area of cutaneous hyperalgesia compared to volunteers treated with placebo, after exposure to the heat/capsaicin model of cutaneous sensitization. Additionally we are going to assess changes in mood/affect and cognitive function of subjects following administration of fenobam and after cutaneous sensitization compared to baseline.

DETAILED DESCRIPTION:
All subjects will receive a topical dose of capsaicin cream 0.1%(Capzasin-HP) to the forearm at the start of the study visit. The order of the 2 treatment regimens indicated below will be randomized and blinded to subjects and researchers.

Treatment Regimen 1: Fenobam [1-(3-chlorophenyl)-3-(1-methyl-4-oxo-2-imidazolidinylidine) urea hydrate]: administration of one 150 mg gelatin capsule.

Treatment Regimen 2: Placebo (lactose monohydrate): administration of one 150 mg gelatin capsule.

ELIGIBILITY:
Inclusion Criteria:

1. 18-50 year old
2. Good general health with no remarkable medical conditions (e.g. liver, kidney, heart, or lung failure)
3. BMI between 20-33
4. Willing to comply with study guidelines as outlined in protocol [including: women of childbearing age must be willing to use a double-barrier method (e.g. oral contraception and condom) for contraception during participation in the study]
5. Willing to provide informed consent

Exclusion Criteria:

1. Anatomical malformation of upper extremities
2. Status post recent trauma or chronic lesions on either forearm
3. Medication use (includes vitamin, herbal, dietary and mineral supplements and grapefruit products during or within 14 days prior to study participation; excludes contraceptives)
4. History of allergy or intolerance to capsaicin
5. History of multiple drug allergies
6. History of addiction to drugs or alcohol (prior or present addiction or treatment for addiction)
7. History of chronic pain syndromes
8. Pregnant and nursing females
9. Smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Suppression of the development of cutaneous hyperalgesia and allodynia around the area treated with heat/capsaicin. | During approximately 7 hours of consecutive assessments
  size of the area of hyperalgesia and allodynia around the area sensitized by heat/capsaicin as quantified by cutaneous stimulation with foam brush strokes and a von Frey filament requiring 26 g of bending force.

SECONDARY OUTCOMES:
Evaluation of nociception after drug administration as evaluated by prolonged (1 min) thermal stimulation on normal (untreated) skin. | During approximately 7 hours of consecutive assessments
  Visual Analog Scale (VAS) rating of pain perception at 1 min 45°C heat stimulation on normal skin.
Assessment of Heat Pain Detection Thresholds (HPDT) in normal and sensitized skin pre and post treatment with fenobam. | During approximately 7 hours of consecutive assessments
  lowest temperature perceived as painful with stimulation starting at 32°C and with a safety cut-off at 52°C.
Absence of significant side effects | 7 days
  Determined by subjects' monitoring during treatment sessions and follow up at 1 day and 1 week after treatment with drug.
Assessment of significant change in mood/affect | During approximately 6 hours of consecutive assessments
  As determined by evaluation of the subjects by combined brief Positive And Negative Affect Scale/Brief State Anxiety Measure (PANAS/BSAM)
Assessment of significant change in cognitive function | During approximately 6 hours of consecutive assessments
  As determined by evaluation of the Letter and Number Sequencing (LNS) assessment

CONTACTS AND LOCATIONS:
Overall Officials: Laura F Cavallone, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States